CLINICAL TRIAL: NCT01424189
Title: Clinical Investigation of AcrySof® IQ ReSTOR® Multifocal Toric Intraocular Lens Models SND1T3/ SND1T4/ SND1T5/ SND1T6
Brief Title: Clinical Investigation of AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric Intraocular Lens (IOL)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C-09-036
Record Dates: First submitted 2011-08-25; First posted 2011-08-26 (Estimated); Results first posted 2017-03-06 (Actual); Last update posted 2018-06-29 (Actual); Status verified 2018-05

CONDITIONS: Cataracts
Keywords: Cataract surgery; Intraocular lens
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ReSTOR Toric IOL (Experimental): AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL, model determined by preoperative keratometric astigmatism, bilateral implantation
  Interventions: Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL
- ReSTOR IOL (Active Comparator): AcrySof® ReSTOR® Multifocal IOL Model SA60D3, bilateral implantation
  Interventions: Device: AcrySof® ReSTOR® Multifocal IOL Model SA60D3

INTERVENTIONS:
Device: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL — Multifocal IOL with extended secondary focal point and astigmatism correction implanted for long-term use over the lifetime of the cataract patient
  Other Names: Models SND1T3, SND1T4, SND1T5, SND1T6
  Arms: ReSTOR Toric IOL
Device: AcrySof® ReSTOR® Multifocal IOL Model SA60D3 — Multifocal IOL with extended secondary focal point implanted for long-term use over the lifetime of the cataract patient
  Arms: ReSTOR IOL

SUMMARY:
The purpose of this study is to evaluate the safety and effectiveness of an investigational multifocal toric intraocular lens (IOL) compared to an FDA-approved multifocal IOL.

DETAILED DESCRIPTION:
Participants 21 years and older within the targeted astigmatism range and in need of cataract extraction in both eyes were consented and randomized in a 2:1 ratio at each investigative site to receive either the AcrySof® IQ ReSTOR® Multifocal Toric IOL or the control AcrySof® ReSTOR® Multifocal IOL in both eyes. Each participant completed a preoperative examination of both eyes, implantation of the IOL at the operative visit for each eye, and up to 8 postoperative visits, with monocular testing at Day 1-2, Day 7-14, and Day 30-60 and binocular testing at Day 120-180 and Day 340-420/Visit 5 following the second implantation. The eye with the greater amount of astigmatism was implanted first (first operative eye). The second eye implant was intended to occur within 30 days after the first eye implant but not prior to 7 days after the first eye implant. Both eyes needed to qualify under inclusion/exclusion criteria at the preoperative visit. If the first eye was excluded during surgery, the second eye was not eligible. If the second eye was excluded during surgery, only the first eye was followed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with bilateral cataracts;
* Able to comprehend and sign a statement of informed consent;
* Calculated lens power and astigmatism within the available range;
* Willing and able to complete all required postoperative visits;
* Planned cataract removal by phacoemulsification;
* Potential postoperative visual acuity of 0.2 logMAR or better in both eyes;
* Preoperative astigmatism in both operative eyes as described in the clinical protocol; Note: Corneal incisions made to reduce astigmatism will not be allowed during the course of the study.
* Clear intraocular media other than cataract in study eyes;
* Preoperative Best Corrected Distance Visual Acuity (BCDVA) worse than 0.2 logMAR in each eye;
* Pupil size greater than or equal to 6 mm after dilation;
* Able to undergo second eye surgery within 30 days of the first eye surgery;
* Other protocol-specified inclusion criteria may apply.

Exclusion Criteria:

* Significant irregular corneal aberration as demonstrated by corneal topography;
* Keratopathy/Kerectasia - any corneal abnormality, other than regular corneal astigmatism;
* Any inflammation or edema (swelling) of the cornea;
* Diagnosed degenerative visual disorders (e.g. macular degeneration or other retinal disorders) that are predicted (by subjective assessment of the retina) to cause future acuity losses to a level worse than 0.2 logMAR;
* Reasonably expected to require a secondary surgical intervention at any time during the study (other than YAG capsulotomy);
* Previous corneal refractive surgery;
* Amblyopia;
* Clinically severe corneal dystrophy (e.g., epithelial, stromal, or endothelial dystrophy);
* Diabetic retinopathy;
* Extremely shallow anterior chamber, not due to swollen cataract;
* Microphthalmos;
* Previous retinal detachment;
* Previous corneal transplant;
* Recurrent severe anterior or posterior segment inflammation of unknown etiology;
* Rubella or traumatic cataract;
* Iris neovascularization;
* Glaucoma (uncontrolled or controlled with medication);
* Aniridia;
* Optic nerve atrophy;
* Pregnancy;
* Current participation in another investigational drug or device study that may confound the results of this investigation;
* Other planned ocular surgery procedures, including, but not limited to LASIK, astigmatic keratotomy and limbal relaxing incisions, for the duration of the study;
* Other protocol-specified exclusion criteria may apply.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 677 (Actual)
Dates: Start 2011-07; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Expert Clinical Project Lead, GCRA, Surgical, Study Director — Alcon Research

REFERENCES:
- [Derived] Williams JR, Kim HW, Crespi CM. Modeling observations with a detection limit using a truncated normal distribution with censoring. BMC Med Res Methodol. 2020 Jun 29;20(1):170. doi: 10.1186/s12874-020-01032-9. PMID 32600261

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 21 investigative sites located in the United States.
Pre-assignment Details: Of the 677 participants enrolled, 103 were exited prior to randomization as screen failures. This reporting population includes all participants with successful IOL implantation in at least 1 eye (574).
Period: Overall Study
Arm/Group | ReSTOR Toric IOL | ReSTOR IOL
Started | 386 | 188
Completed | 373 | 182
Not Completed | 13 | 6
Not completed — Adverse Event | 1 | 0
Not completed — Lost to Follow-up | 4 | 1
Not completed — Withdrawal by Subject | 4 | 4
Not completed — Subject moved | 1 | 0
Not completed — Death | 3 | 1

BASELINE CHARACTERISTICS:
Population: This analysis population includes all participants with successful IOL implantation in at least 1 eye.
Groups:
- Total: Total of all reporting groups
Arm/Group | ReSTOR Toric IOL | ReSTOR IOL | Total
Number analyzed (Participants) | 386 | 188 | 574
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.91 (9.20) | 68.36 (8.13) | 67.38 (8.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 240 | 136 | 376
  Male | 146 | 52 | 198

OUTCOME MEASURES:

1. Primary Outcome: Mean Monocular Uncorrected Distance Visual Acuity (UCDVA) at Fixed Distance at Visit 5
Description: Visual acuity (VA) was measured monocularly (each eye separately) without visual correction using a 100% contrast ETDRS (Early Treatment of Diabetic Retinopathy Study) chart positioned 4 meters (m) from the participant under well-lit conditions. +0.25 diopter (D) spherical power was applied to correct for optical infinity. VA was measured in logMAR (logarithm of the minimum angle of resolution), with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity. This analysis was prespecified for the first operative eye.
Time Frame: Month 12 from second eye implantation
Population: This analysis population includes all participants with successful IOL implantation in the first implanted eye with data at visit.
Measure: Least Squares Mean (Standard Error); unit: logMAR
Units Other Than Participants: eyes
Groups:
- ReSTOR Toric IOL: AcrySof® IQ ReSTOR® +3.0 D Multifocal Toric IOL, model determined by preoperative keratometric astigmatism
- ReSTOR IOL: AcrySof® ReSTOR® Multifocal IOL Model SA60D3
Arm/Group | ReSTOR Toric IOL | ReSTOR IOL
Number analyzed (Participants) | 373 | 180
Number analyzed (eyes) | 373 | 180
logMAR | 0.126 (0.013) | 0.125 (0.015)
Statistical Analysis 1: Comparison: ReSTOR Toric IOL vs ReSTOR IOL; Test type: Non-Inferiority or Equivalence — With 300 subjects in the ReSTOR Toric IOL test group and 150 subjects in the ReSTOR IOL control group, there was over 99% power to demonstrate that the upper 95% confidence limit for the observed difference in UCDVA between IOL groups was less than the clinical performance target of 0.1 logMAR units at Month 12, assuming the true difference between groups is zero. This was based on an assumed standard deviation for UCDVA of 0.16 logMAR units and a 1-sided, α=0.05 test; Mean Difference (Final Values) = 0.001, 95% CI 1-sided [upper limit 0.030], Standard Error of Mean 0.013

2. Primary Outcome: Mean Monocular Uncorrected Near Visual Acuity (UCNVA) at Fixed Distance at Visit 5
Description: VA was measured monocularly without visual correction using a hand-held ETDRS chart at a fixed distance that differed by lens model implanted. The logMAR ETDRS near visual acuity chart was designed for use at 40 cm; results obtained at other distances were converted to reflect the change in apparent letter size that results from the change in distance. VA was measured in logMAR, with 0.1 logMAR increment corresponding to 5 letters, or 1 line, on an ETDRS chart. A lower numeric value represents better visual acuity. This analysis was prespecified for the first operative eye.
Time Frame: Month 12 from second eye implantation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: logMAR
Arm/Group | ReSTOR Toric IOL | ReSTOR IOL
Number analyzed (Participants) | 373 | 180
logMAR | 0.19 (0.015) | 0.24 (0.017)
Statistical Analysis 1: Comparison: ReSTOR Toric IOL vs ReSTOR IOL; Test type: Non-Inferiority or Equivalence — With 300 subjects in the ReSTOR Toric IOL test group and 150 subjects in the ReSTOR IOL control group, there was over 99% power to demonstrate that the upper 95% confidence limit for the observed difference in UCNVA between IOL groups was less than the clinical performance target of 0.1 logMAR units at Month 12, assuming the true difference between groups is zero. This estimate was based on an assumed standard deviation for UCNVA of 0.16 logMAR units and a 1-sided, α=0.05 test; Mean Difference (Final Values) = -0.044, 95% CI 1-sided [upper limit -0.017], Standard Error of Mean 0.015

3. Primary Outcome: Rate of Actual and Potential Secondary Surgical Interventions (SSIs) Related to the Optical Properties of the IOL for First and Second Operative Eyes Separately at Visit 5
Description: The rate of actual and potential secondary surgical interventions (SSIs) related to the optical properties of the IOL was estimated. If an ocular surgical intervention was performed, it qualified as an actual SSI; however; if the participant met the protocol-specified criteria that would warrant an SSI, but didn't actually undergo the SSI, it qualified as a potential SSI. Rate is presented as percentage of participants.
Time Frame: Month 12 from second eye implantation
Population: This analysis population includes all participants with attempted IOL implantation (successful or aborted after contact with the eye). For participants with actual SSIs, performance testing outcomes conducted prior to the secondary intervention were carried forward to the final analysis.
Measure: Number; unit: percentage of participants
Arm/Group | ReSTOR Toric IOL | ReSTOR IOL
Number analyzed (Participants) | 386 | 188
percentage of participants
  First Implanted Eye | 1.04 | 2.13
  Second Implanted Eye: number analyzed (Participants) | 383 | 188
  Second Implanted Eye | 0.52 | 2.13

4. Secondary Outcome: Rate of Severe Visual Disturbances/Distortions Reported on the Assessment of Photic Phenomena & Lens EffectS (APPLES) Questionnaire at Visit 5
Description: Visual disturbances/distortions were reported by the participant on the Assessment of Photic Phenomena and Lens EffectS (APPLES) questionnaire, a Patient Reported Outcome (PRO) questionnaire intended to evaluate 10 distinct visual phenomena associated with cataract extraction and IOL implantation. The first 20 questions addressed both the frequency and severity of the phenomena using a 4-point categorical scale ranging from "never" to "always" (frequency) or "none" to "severe" (severity). The final (21st) question indicated whether the participant answered the questions based on experiences with or without glasses. The participant completed the assessment as a retrospective analysis of the previous week. Rate is presented as the percentage of participants with severity score "severe" for the visual phenomenon.
Time Frame: Month 12 from second eye implantation
Population: This analysis population includes all participants with attempted IOL implantation (successful or aborted after contact with the eye).
Measure: Number; unit: percentage of participants
Arm/Group | ReSTOR Toric IOL | ReSTOR IOL
Number analyzed (Participants) | 386 | 188
percentage of participants
  Blurred vision: number analyzed (Participants) | 372 | 182
  Blurred vision | 0.8 | 0.0
  Color distortion: number analyzed (Participants) | 371 | 182
  Color distortion | 0.0 | 0.0
  Flat lines look curved: number analyzed (Participants) | 372 | 182
  Flat lines look curved | 0.0 | 0.0
  Straight lines look tilted: number analyzed (Participants) | 372 | 182
  Straight lines look tilted | 0.0 | 0.0
  Double vision: number analyzed (Participants) | 372 | 182
  Double vision | 0.8 | 0.0
  Feeling sick due to visual distortion: number analyzed (Participants) | 371 | 182
  Feeling sick due to visual distortion | 0.0 | 0.5
  Glare: number analyzed (Participants) | 372 | 182
  Glare | 3.5 | 2.7
  Halos: number analyzed (Participants) | 372 | 182
  Halos | 7.5 | 11.0
  Hazy vision: number analyzed (Participants) | 372 | 182
  Hazy vision | 1.3 | 0.5
  Starbursts: number analyzed (Participants) | 372 | 182
  Starbursts | 4.3 | 8.8

ADVERSE EVENTS:
Time Frame: This analysis group includes all participants with attempted IOL implantation (successful or aborted after contact with the eye).
Description: An Adverse Event (AE) was defined as any untoward medical occurrence, unintended disease or injury, or untoward clinical sign, whether or not related to the investigational device. AEs were collected as solicited comments and as observations by the Investigator as outlined in the protocol. "At Risk" population for ocular AEs is included with unit of "eyes."
Arm/Group | ReSTOR Toric IOL | ReSTOR IOL
Serious Adverse Events (participants affected / at risk) | 45/386 | 21/188
Other Adverse Events (participants affected / at risk) | 48/386 | 28/188
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ReSTOR Toric IOL (N=386) | ReSTOR IOL (N=188)
Atrial fibrillation (Cardiac disorders) | 1 | 1
Bradycardia (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 0 | 1
Coronary artery disease (Cardiac disorders) | 0 | 2
Age-related macular degeneration (First Implanted Eye) (Eye disorders) | 0 | 1
Cystoid macular oedema (First Implanted Eye) (Eye disorders) | 1 | 0
Cystoid macular oedema (Second Implanted Eye) (Eye disorders) | 3/383 | 1
Eye disorder (First Implanted Eye) (Eye disorders) | 1 | 0
Eye disorder (Second Implanted Eye) (Eye disorders) | 3/383 | 0
Glare (First Implanted Eye) (Eye disorders) | 1 | 0
Glare (Second Implanted Eye) (Eye disorders) | 1/383 | 0
Halo vision (First Implanted Eye) (Eye disorders) | 1 | 1
Halo vision (Second Implanted Eye) (Eye disorders) | 1/383 | 2
Iris atrophy (First Implanted Eye) (Eye disorders) | 1 | 0
Iris atrophy (Second Implanted Eye) (Eye disorders) | 1/383 | 0
Macular hole (Second Implanted Eye) (Eye disorders) | 1/383 | 0
Macular oedema (Second Implanted Eye) (Eye disorders) | 0/383 | 1
Photopsia (First Implanted Eye) (Eye disorders) | 1 | 0
Photopsia (Second Implanted Eye) (Eye disorders) | 1/383 | 0
Retinal detachment (First Implanted Eye) (Eye disorders) | 1 | 0
Retinal detachment (Second Implanted Eye) (Eye disorders) | 2/383 | 1
Retinal tear (Second Implanted Eye) (Eye disorders) | 1/383 | 0
Vision blurred (First Implanted Eye) (Eye disorders) | 1 | 0
Vision blurred (Second Implanted Eye) (Eye disorders) | 0/383 | 1
Visual impairment (First Implanted Eye) (Eye disorders) | 1 | 1
Visual impairment (Second Implanted Eye) (Eye disorders) | 1/383 | 1
Vitreous prolapse (First Implanted Eye) (Eye disorders) | 1 | 0
Colitis (Gastrointestinal disorders) | 1 | 0
Colitis ischaemic (Gastrointestinal disorders) | 0 | 1
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 | 0
Hiatus hernia (Gastrointestinal disorders) | 1 | 0
Peptic ulcer (Gastrointestinal disorders) | 2 | 0
Death (General disorders) | 1 | 0
Device dislocation (First Implanted Eye) (General disorders) | 1 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Cholecystitis chronic (Hepatobiliary disorders) | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0
Pyothorax (Infections and infestations) | 1 | 0
Sepsis (Infections and infestations) | 1 | 0
Cataract operation complication (First Implanted Eye) (Injury, poisoning and procedural complications) | 2 | 0
Cataract operation complication (Second Implanted Eye) (Injury, poisoning and procedural complications) | 1/383 | 1
Eye injury (Second Implanted Eye) (Injury, poisoning and procedural complications) | 1/383 | 0
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Surgical procedure repeated (First Implanted Eye) (Injury, poisoning and procedural complications) | 3 | 2
Surgical procedure repeated (Second Implanted Eye) (Injury, poisoning and procedural complications) | 1/383 | 3
Wound complication (Second Implanted Eye) (Injury, poisoning and procedural complications) | 1/383 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Breast cancer stage III (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Gastric neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dementia (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0
Mental status changes (Psychiatric disorders) | 1 | 0
Renal failure acute (Renal and urinary disorders) | 2 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Non-cardiogenic pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cholecystectomy (Surgical and medical procedures) | 0 | 1
Corneal operation (First Implanted Eye) (Surgical and medical procedures) | 1 | 1
Corneal operation (Second Implanted Eye) (Surgical and medical procedures) | 1/383 | 1
Eye laser surgery (First Implanted Eye) (Surgical and medical procedures) | 1 | 0
Eye laser surgery (Second Implanted Eye) (Surgical and medical procedures) | 3/383 | 0
Intraocular injection (First Implanted Eye) (Surgical and medical procedures) | 0 | 1
Intraocular lens repositioning (First Implanted Eye) (Surgical and medical procedures) | 4 | 0
Keratometry (First Implanted Eye) (Surgical and medical procedures) | 1 | 0
Keratomileusis (First Implanted Eye) (Surgical and medical procedures) | 1 | 0
Keratomileusis (Second Implanted Eye) A (Surgical and medical procedures) | 1/383 | 0
Knee arthroplasty (Surgical and medical procedures) | 1 | 0
Retinal operation (Second Implanted Eye) (Surgical and medical procedures) | 1/383 | 0
Retinopexy (First Implanted Eye) (Surgical and medical procedures) | 2 | 0
Retinopexy (Second Implanted Eye) (Surgical and medical procedures) | 3/383 | 1
Rotator cuff repair (Surgical and medical procedures) | 1 | 0
Suture insertion (Second Implanted Eye) (Surgical and medical procedures) | 1/383 | 1
Vitrectomy (First Implanted Eye) (Surgical and medical procedures) | 1 | 0
Aortic stenosis (Vascular disorders) | 1 | 0
Orthostatic hypotension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | ReSTOR Toric IOL (N=386) | ReSTOR IOL (N=188)
Dry Eye (Second Implanted Eye) (Eye disorders) | 8/383 | 10
Posterior capsule opacification (First Implanted Eye) (Eye disorders) | 35 | 17
Posterior capsule opacification (Second Implanted Eye) (Eye disorders) | 32/383 | 19

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.